CLINICAL TRIAL: NCT00694291
Title: Phase II Double Blind Randomized Placebo Controlled Study of Sorafenib in Hormone Naïve Biochemical Recurrence of Prostate Cancer
Brief Title: Sorafenib in Hormone Naïve Biochemical Recurrence of Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Yu-Ning Wong MD, Associate Member, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FCCC 07-038
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Prostate Cancer
Keywords: Rising PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sorafenib 400 mg orally twice daily
  Interventions: Drug: Sorafenib
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sorafenib — 400 mg orally twice daily
  Other Names: Nexavar
  Arms: 1
Drug: Placebo — Matching Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to measure the benefit of sorafenib in patients with a rising PSA after treatment with radiation therapy or surgery who are NOT receiving with androgen ablation therapy.

DETAILED DESCRIPTION:
This is a placebo controlled double blind study of sorafenib versus placebo of in patients with high risk biochemical recurrence of prostate cancer. High risk characteristics include a short PSADT (<9 months) or high Gleason score (>8), characteristics, which correspond to a higher risk of prostate cancer specific mortality in patients with biochemical recurrence following radiation therapy or radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Prior definitive treatment with radical prostatectomy and/or radiation therapy (external beam or brachytherapy). Patients may have received post prostatectomy radiation therapy in the adjuvant setting or for biochemical recurrence.
* Hormone sensitive prostate cancer as evidence by a serum total testosterone level within the institution's normal range £4 weeks of registration. (Patients may have received hormonal therapy in the adjuvant setting provided the last dose was ³ one year from the date of enrollment.)
* All patients must have evidence of biochemical progression as determined by 3 PSA measures. (PSA-2, PSA-1 and PSA 0) The most recent PSA value (PSA0) will serve as the baseline. All of these PSA values must be obtained at the same reference lab and the earliest (PSA-2) ≥ eight weeks prior to registration, but ≤ six months prior to enrollment.
* The most recent PSA value (PSA 0) must be drawn £ seven days of treatment and must be greater than 0.4 ng/ml (after prostatectomy) or greater than ³1.5 ng ml (after radiation therapy) at the time of registration.
* The patient must be at high risk for developing distant metastases by one of the following criteria:

  * Gleason score 8-10 on original tumor specimen or
  * Prostate specific antigen doubling time (PSADT) less than nine months calculated using the following formula PSADT in days = 0.693 (t) ln( PSA-1)-ln (PSA-2)

where t = number of days between PSA- 2 and PSA-1 PSA-1 is the most recent PSA value PSA-2 is the next most recent PSA value Ln = natural log PSADT in months = PSADT divided by 30.4

* Age > 18 years old
* ECOG Performance Status 0 or 1
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin > 9.0 g/dl
  * Absolute neutrophil count (ANC) > 1,500/mm3
  * Platelet count > 100,000/mm3
  * Total bilirubin < 1.5 times ULN
  * ALT and AST < 2.5 times the ULN
  * Creatinine < 1.5 times ULN
  * INR < 1.5 or a PT/PTT within normal limits in patients not on therapeutic anticoagulation. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of Sorafenib and monitored at least weekly, or as defined by the local standard of care, until INR is stable.
* Men should agree to use adequate birth control during and for at least three months after the last administration of Sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
* Consideration must be given to definitive local therapy; patient may either refuse or not be considered a candidate.

Exclusion Criteria:

* Therapy modulating testosterone levels (such as leuteinizing-hormone releasing hormone agonists/antagonists and antiandrogens) for treatment of biochemical recurrence of prostate cancer. Treatment in the neoadjuvant setting is permissible if greater than 1 year prior to registration. Agents such as 5 alpha reductase inhibitors, ketoconazole, megestrol acetate, systemic steroids, or herbal supplements that are known to affect PSA (PC Spes, saw palmetto oil) are not permitted at any time during the period that the PSA values are being collected during screening or treatment
* Evidence of measurable or evaluable metastatic disease on chest x-ray bone scan or CT scan performed ≤ four weeks of registration.
* Patients must not have received any other investigational agents or concurrent anti cancer therapy £4 weeks from treatment.
* Cardiac disease: Congestive heart failure > class II NYHA. Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began ≤ the last 3 months) or myocardial infarction ≤ the past 6 months.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Sorafenib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies may be undertaken in patients receiving combination antiretroviral therapy in the future
* Active clinically serious infection > CTCAE Grade 2.
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks ≤ the past 6 months.
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 £4 weeks of registration.
* Any other hemorrhage/bleeding event >CTCAE Grade 3 £ 4 weeks of registration.
* Evidence or history of bleeding diathesis or coagulopathy
* Major surgery, open biopsy or significant traumatic injury ≤ 4 weeks of registration.
* Concurrent use of cytochrome P450 enzyme inducing antiepileptic drugs (phenytoin, carbamazepine, and phenobarbital), rifampin or St Johns Wort. Patients must have discontinued these medications ³14 days from starting protocol therapy
* Known or suspected allergy to Sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.
* Any malabsorption problem.
* Prior history of cancer (except basal cell or squamous cell skin cancer) ≤ the past five years.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To compare the median PSA slope of patients with non-castrate, high risk biochemical recurrence of prostate cancer following definitive local therapy treated with Sorafenib for six months compared to those treated with placebo. | 6 months

SECONDARY OUTCOMES:
To determine the response rate based on PSA criteria and duration of PSA response. | 6 months
To compare the time to PSA progression between the Sorafenib arm and the placebo arm. | 6 months
To document the safety and tolerability of Sorafenib in this patient population. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ning Wong, MD MSCE, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States